CLINICAL TRIAL: NCT03679650
Title: A Phase I Clinical Trial of Dendritic Cell/AML Fusion Cell Vaccine Alone and in Conjunction With Decitabine Following Allogeneic Transplantation in AML Patients
Brief Title: Dendritic Cell/AML Fusion Cell Vaccine Following Allogeneic Transplantation in AML Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jacalyn Rosenblatt, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-202; 1P50CA206963-01A1 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AML Patient who are undergoing allogeneic transplantation (Experimental): * Patients will be vaccinated with DC/AML fusion cells
  * Four days of GM-CSF given subcutaneously at the site of vaccination
  * Patients will receive 2 vaccines, 3 weeks apart, with the potential for a booster vaccine
  * Patients will be treated with 5 days of decitabine in the post-transplant setting
  Interventions: Biological: DC/AML fusion cells
- AML Patient who are undergoing transplantation (Experimental): * Patients will be vaccinated with DC/AML fusion cells
  * Four days of GM-CSF given subcutaneously at the site of vaccination
  * Patients will receive 2 vaccines, 3 weeks apart, with the potential for a booster vaccine
  Interventions: Biological: DC/AML fusion cells

INTERVENTIONS:
Biological: DC/AML fusion cells — An investigational agent that tries to help the immune system to recognize and fight against cancer cells

SUMMARY:
This research study is studying a cancer vaccine called Dendritic Cell/AML Fusion vaccine (DC/AML vaccine) as a possible treatment for Acute Myelogenous Leukemia (AML).

The interventions involved in this study are:

* Dendritic Cell/AML Fusion vaccine (DC/AML vaccine)
* Decitabine, a chemotherapy drug

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. This study is investigating the DC/AML vaccine with and without the drug decitabine as a possible treatment for AML in the post-transplant setting.

The FDA (the U.S. Food and Drug Administration) has not approved the DC/AML vaccine as a treatment for any disease.

The FDA has approved decitabine as a treatment option for this disease.

The FDA has not approved the combination of the DC/AML vaccine with decitabine as a treatment option for any disease,

In this research study, the investigators are determining if the DC/AML vaccine can be used safely in subjects with acute leukemia after they have undergone a transplant, and whether the DC/AML vaccine alone is capable of producing immune responses against leukemia. Cancer cells are foreign to the body and have unique markers that distinguish them from normal cells.

These markers can potentially serve as targets for the immune system. An immune response is any reaction by the immune system; a complex system that is responsible for distinguishing us from everything foreign to us, and for protecting us against infections and foreign substances.

The DC/AML vaccine is an investigational agent that tries to help the immune system to recognize and fight against cancer cells. Unlike a standard vaccine that is used to prevent infections, cancer vaccines are being studied to see if they can fight cancers that are already in the body. Laboratory studies have shown that when dendritic cells and tumor cells are brought together, the dendritic cells can stimulate immune responses against the tumor and, in some cases, cause the tumor to shrink.

Decitabine is thought to act as an anti-metabolite. It seems to work by having a toxic effect on the abnormal bone marrow cells. It also appears to affect the DNA in genes that control cell growth. This promotes normal specialization and blood cell growth, so that the body is better able to make red blood cells, white blood cells, and platelets.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML who have undergone AML cell harvest and cryopreservation as per protocol 16-593 or companion protocol 18-232.
* Patients must have had a minimum of 5x107 cells cryopreserved.
* Patients must be day 25-45 following allogeneic transplantation from either:

  * Group A: HLA 8/8 or 7/8 matched related donor or HLA 8/8 matched unrelated donor, as determined by antigen or allele level typing at HLA A,B,C, and HLA DRB1.

OR

* Group B: Haplo-identical donor

  * Patients must be ≥ 18 years old
  * ECOG performance status ≤2 (Appendix A)
  * Participants must have normal organ and marrow function as defined below:
* Total bilirubin ≤ 2.0 mg/dL (unless patient has Gilbert's disease)
* AST(SGOT)/ALT(SGPT) ≤ 3 × institutional upper limit of normal
* Creatinine ≤ 2.0 mg/dl
* Absolute neutrophil count > 1000
* Platelet count > 50,000

  * The effects of DC/AML fusion cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  * No evidence of ongoing grade 2 or higher aGVHD
  * Must be on prednisone <20mg or other steroid equivalent
  * Donor chimerism of bone marrow >60%
  * Resolution of all transplant related grade III-IV toxicity as per CTC criteria 4.0
  * Complete remission defined by absence of circulating blasts and less than 5% blasts in the bone marrow
  * Ability to understand and the willingness to sign a written informed consent document.

Eligibility Prior to Initiating Vaccination (Groups A and B)

* Assessments to be done between Day 45-75 post-transplant.
* At least 2 doses of fusion vaccine were produced
* No ongoing grade II-IV acute GVHD
* Prednisone requirement of < 20mg a day or steroid equivalent
* Participants must have normal organ and marrow function as defined below:

  * Total bilirubin ≤ 2.0 mg/dL (unless patient has Gilbert's disease)
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional upper limit of normal
  * Creatinine ≤ 2.0 mg/dl
  * Absolute neutrophil count > 1000
  * Platelet count > 50,000
* No uncontrolled acute infection
* No CTCAE grade ≥ 3 non-hematologic toxicity
* No serious intercurrent illness such as active acute infection, or significant cardiac disease characterized by clinically significant arrhythmia, active ischemic coronary disease or symptomatic congestive heart failure.
* Participants must be in a complete remission

Pre-Treatment Criteria Prior to Decitabine (Group A Cohort 2)

* Assessments to be done within 3 days prior to initiation of therapy.
* Participants must have normal organ and marrow function as defined below:
* Total bilirubin ≤ 2.0 mg/dL (unless patient has Gilbert's disease)

  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional upper limit of normal
  * Creatinine ≤ 2.0 mg/dl
  * Absolute neutrophil count > 1000
  * Platelet count > 50,000

Exclusion Criteria:

* Because of compromised cellular immunity, patients with a known history of HIV are excluded
* Leukemia with active CNS involvement
* Patients must not be pregnant. All premenopausal patients will undergo pregnancy testing. Men will agree to not father a child while on protocol treatment. Men and women will practice effective birth control while receiving protocol treatment.
* Participants may not be receiving any other Non-FDA approved study agents at the start of vaccination
* Uncontrolled intercurrent illness including uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements.
* Autoimmune or inflammatory disorders requiring active treatment with systemic steroids or immunosuppressive therapy limited to the following:

  * GI Disorders: (including inflammatory bowel disease [e.g., ulcerative colitis, Crohn's disease]
  * Systemic lupus erythematosus
  * Wegener's syndrome [granulomatosis with polyangiitis]
  * Myasthenia gravis
  * Graves' disease
  * Rheumatoid arthritis
  * Hypophysitis
  * Uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The fold-increase in AML specific T cells in peripheral blood and bone marrow | 12 months
  The fold-increase in AML specific T cells in the peripheral blood and bone marrow

SECONDARY OUTCOMES:
Complete Remission | 12 months
  Patients in complete remission
Complete Remission with Incomplete Count Recovery | 12 Months
  Patients in complete remission with incomplete count recovery
Complete Remission with Incomplete Platelet Recovery | 12 months
  Patients in complete remission with incomplete platelet recovery
Partial Remission (PR) | 12 months
  Patients in Partial Remission
Rate of Relapse | 12 months
  Rate of relapse seen in patients
Stable Disease | 12 Months
  Patients with stable disease
Relapse free survival | 12 Months
  Patients with relapse free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No